CLINICAL TRIAL: NCT02383732
Title: A Feasibility Study of the Elopement Prevention and Safety Training Program
Brief Title: A Study of the Elopement Prevention and Safety Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nathan A. Call, Ph.D., BCBA-D, Instructor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00076337
Record Dates: First submitted 2015-02-25; First posted 2015-03-09 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Elopement; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Pediatric subjects between the age of 4-12 years with autistic spectrum disorder and elopement will begin the Elopement Prevention and Safety Training (EPST) program. EPST includes up to 12 120-minute weekly sessions delivered over approximately 12-14 weeks. EPST is a modular treatment, with three components: 1) Universal Safety Measures (USM), 2) Proximity training, and 3) Check-in training. All participants receive the USM module in the first two sessions. They then receive either the Proximity training or Check-in training module depending on the type of elopement exhibited by the child (i.e., bolting vs. wandering).
  Interventions: Behavioral: Universal Safety Measures Module (All participants); Behavioral: Proximity Training Module (Bolting Prevention Participants); Behavioral: Check-In Training Module (Wandering Prevention Participants)
- Waitlist Control (Active Comparator): Pediatric subjects between the age of 4-12 years with autistic spectrum disorder and elopement will be assigned to the Waitlist Control group. The subjects will be offered the intervention after completion of the 12-week waiting period. The subjects will then begin the Elopement Prevention and Safety Training (EPST) program. EPST includes up to 12 120-minute weekly sessions delivered over approximately 12-14 weeks. EPST is a modular treatment, with three components: 1) Universal Safety Measures (USM), 2) Proximity training, and 3) Check-in training. All participants receive the USM module in the first two sessions. They then receive either the Proximity training or Check-in training module depending on the type of elopement exhibited by the child (i.e., bolting vs. wandering).
  Interventions: Behavioral: Universal Safety Measures Module (All participants); Behavioral: Proximity Training Module (Bolting Prevention Participants); Behavioral: Check-In Training Module (Wandering Prevention Participants)

INTERVENTIONS:
Behavioral: Universal Safety Measures Module (All participants) — During the first session, the therapist conducts a home safety evaluation. During the second visit the therapist provides the caregiver with an individualized Elopement Prevention & Safety Plan (EPSP) based upon the results of the evaluation. The remainder of the session is spent helping caregivers make plans to implement the EPSP to reduce the risk of elopement or lessen the risk of harm to the child if they do successfully elope.
Behavioral: Proximity Training Module (Bolting Prevention Participants) — During the first session a functional behavioral assessment (FBA) of bolting is conducted to identify the motivator(s) that evoke bolting. Caregivers identify a setting that is most problematic because it contains the item/activity that most frequently serves as a motivator for elopement. In the next session, caregivers are taught to identify effective alternative reinforcers. In subsequent sessions, antecedent and consequence based strategies are employed to reduce motivation for elopement and reinforce remaining within the designated proximity of a caregiver for increasing durations.
Behavioral: Check-In Training Module (Wandering Prevention Participants) — This module employs behavioral strategies to teach a child to check in with a caregiver at frequent fixed intervals during periods of low supervision. Delivering potent reinforcement for checking in counteracts any motivation to wander. Furthermore, if the child does wander caregivers become aware of it immediately because they failed to check in. During the first session caregivers are taught to identify effective reinforcers. A vibrating alarm that can be carried in a participating child's pocket serves as a prompt to seek out a caregiver and check-in. Participants receive access to a previously identified and individualized reinforcer for checking-in with the caregiver.

SUMMARY:
The purpose of this study is to demonstrate the feasibility of the Elopement Prevention Safety (EPST) program in children with autism spectrum disorder (ASD) who have engaged in eloping. This is a program created by the Behavior Treatment Clinics to help caregivers come up with a safety plan to prevent their children from running away or wandering off.

DETAILED DESCRIPTION:
A large number of children with autism spectrum disorder (ASD) have a current or past history of elopement. For parents of a child with ASD, having their child go missing is potentially dangerous and far more likely compared to typically developing children. This behavior interferes with household routines, engenders vigilance, and restricts the family's participation in their community. Such restrictions contribute to the family's isolation and hinders development of community supports. Elopement can result in injuries and deaths of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 4 to 12 inclusive
2. Diagnosis of ASD as determined by clinical interview and supported by standardized measures (i.e., Autism Diagnostic Observation Schedule-2, Vineland, Stanford-Binet V)
3. Engages in elopement in the form of bolting or wandering, as determined by structured interview
4. A caregiver who expresses a willingness to participate in treatment and complete baseline/outcome assessments.

Exclusion Criteria:

1. Unmanaged psychopathology or problem behavior other than elopement that warrants immediate clinical care, determined by clinical interview and Aberrant Behavior Checklist (ABC)
2. Child and family currently in therapy that is likely to be redundant with the treatment program or interfere with proposed treatment
3. Presence of both of the types of elopement under investigation (i.e., both bolting and wandering).

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention, assessed by change in severity on Clinical Global Impression for Severity (CGI-S) | Post-intervention (12-14 weeks)
  An independent evaluator (IE) will conduct a parent target problem survey to help caregivers estimate the frequency of elopement as well as its impact on the family. From this description, the IE (who will be blind to treatment assignment) will generate a brief narrative describing the participant's elopement. This narrative will be used by the IE to rate the overall severity on the 7-point Clinical Global Impression for Severity (CGI-S). Clinical Global Impression of Severity (CGI-S) Scale is a clinician's assessment of patient's severity of illness. The score ranges from 1 = normal, not at all ill to 7 = among the most extremely ill patients

SECONDARY OUTCOMES:
Change in elopement behavior | Post-intervention (12-14 weeks)
  Number of times a subject exhibits bolting and wandering at baseline and post-intervention. Change in elopement will be subtracting the number of bolting and wandering events from post-intervention and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Call, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Lomas Mevers J, Call NA, Gerencser KR, Scheithauer M, Miller SJ, Muething C, Hewett S, McCracken C, Scahill L, McElhanon BO. A Pilot Randomized Clinical Trial of a Multidisciplinary Intervention for Encopresis in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2020 Mar;50(3):757-765. doi: 10.1007/s10803-019-04305-5. PMID 31768718